CLINICAL TRIAL: NCT05826873
Title: Implementing a Discharge Stewardship Bundle to Improve Antibiotic Use at Transition From Hospital to Home
Brief Title: Discharge Stewardship in Children's Hospitals
Acronym: DISCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Seattle Children's Hospital (Other); Primary Children's Hospital (Other); St. Louis Children's Hospital (Other); University of Pennsylvania (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-017269; R01HS027428-01 (AHRQ)
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia, Bacterial; Pneumonia Childhood; Urinary Tract Infections; Soft Tissue Infections; Skin Infections; Community-acquired Pneumonia
Keywords: Stewardship; Discharge Stewardship; Group-level feedback; Antibiotic; Community-acquired pneumonia; Skin and soft tissue infections; Urinary Tract Infections
MeSH Terms: conditions — Pneumonia, Bacterial; Urinary Tract Infections; Soft Tissue Infections; Cellulitis; Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Mixed methods implementation science study with a multicenter, quasi-experimental interrupted time-series design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Hospitalists (Other): Prescribing physicians and hospital employees will be recruited during regularly held staff meetings prior to the data collection period. The study team will briefly introduce the study aims and methods and let the hospitalists know that the study team will be emailing them separately to ask permission for Dr. Szymczak to shadow them. Only those who have agreed will participate in the ethnographic observations. For the interviews and surveys, the study team will recruit respondents via contact made during ethnographic observations. The study team will also utilize a snowball approach by asking respondents if they know of any other staff who might be interested in participating in an interview. Approximately 120 clinicians will participate in the interviews and surveys.
  Interventions: Behavioral: Discharge antibiotic stewardship intervention
- Families of hospitalized children (No Intervention): Families of children who were hospitalized at one of the four participating sites will be approached for consent to participate in the study. Families who consent will complete 2 brief REDCap surveys and a wellness tracker after their child is discharged from the hospital.

INTERVENTIONS:
Behavioral: Discharge antibiotic stewardship intervention — Hospitalists will be provided with group-level, quarterly feedback reports illustrating the number of prescriptions that had the appropriate antibiotic duration and appropriate antibiotic choice for each of the three conditions.
  Arms: Pediatric Hospitalists

SUMMARY:
The goal of this interventional study is to test if a discharge stewardship bundle is effective at reducing inappropriate antibiotic prescriptions at hospital discharge for children with the three common infections: community-acquired pneumonia (CAP), urinary tract infections (UTI), and skin/soft tissue infections (SSTI). The goals of this study are:

* To develop, locally adapt, and implement a discharge stewardship intervention across four geographically diverse children's hospitals.
* To measure the impact of the discharge stewardship intervention on antibiotic prescribing and patient outcome for three common pediatric infections.

Families who are enrolled in the study will be asked to:

* complete a one question wellness track on days 3, 7, and 21 after hospital discharge
* complete a brief survey on days 7 and 21 after hospital discharge

The study team will conduct interviews with the hospitalists at each of the four participating hospitals to create a "discharge stewardship" bundle. Once the bundle intervention is implemented, the hospitalists will be asked to follow prescribing guidelines for CAP, UTI, and SSTI. They will receive regular group-level feedback reports to show how well they follow the guidelines and motivate the hospitalists to follow the guidelines better.

DETAILED DESCRIPTION:
Pediatric antibiotic stewardship programs (ASPs) in hospital and outpatient settings optimize the use of antibiotics to improve clinical outcomes, decrease adverse drug events, and reduce the emergence of antibiotic resistant bacteria. However, stewardship for patients at the transition from hospital discharge to home, or "discharge stewardship," is an unmet need for several reasons. First, few pediatric stewardship programs perform discharge stewardship. Second, approximately 30% of pediatric patients receive antibiotics at hospital discharge. Third, the majority of antibiotic days prescribed for hospitalized patients occur after discharge. Fourth, up to half of discharge antibiotic prescriptions are suboptimal, which includes choosing the wrong drug, dose, route, or duration of therapy.

This project will use an implementation science framework to develop, implement, and test the effectiveness of a multifaceted discharge stewardship intervention for hospitalized children with the three most common indications for antibiotic prescribing in hospitalized children - community acquired pneumonia (CAP), urinary tract infections (UTI), and skin/soft tissue infections (SSTI) - at four children's hospitals to establish a foundation for future expansion to additional target populations. Antibiotic choice, dose, route, and duration of therapy will be addressed.

Aim 1 is to develop, locally adapt, and implement a discharge stewardship intervention across the four participating sites. The integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework will guide a rapid formative evaluation to identify contextual factors likely to facilitate or hinder the implementation of a discharge stewardship intervention at each site. Based on these results, local facilitators will work to develop and implement a discharge stewardship intervention comprised of consensus driven clinical prescribing guidelines for CAP, UTI, and SSTI plus quarterly feedback of prescribing data based on these guidelines. Aim 2 is to measure the impact of the discharge stewardship intervention on antibiotic prescribing (the primary outcome) and patient-centered balancing measures (post-discharge treatment failure and adverse events).

This project will form the foundation for future dissemination of discharge stewardship to a broader array of patient populations. Investigators on this proposal form the leadership of the Sharing Antimicrobial Reports for Pediatric Stewardship (SHARPS) Collaborative, a network comprised of more than 60 children's hospitals across North America that is uniquely positioned to adopt antimicrobial stewardship interventions designed to target prescribing at hospital discharge.

ELIGIBILITY:
Clinician Inclusion Criteria

1. >18 year old
2. Employed by the hospital as an attending physician, advanced practice provider, resident trainee or other clinical stakeholder (e.g. pharmacist, infectious diseases attending)

Clinician Exclusion Criteria

1. <18 years old
2. Not employed by the hospital

Patient Inclusion Criteria

1. Subjects less than 18 years
2. Diagnosed with either uncomplicated community acquired pneumonia, urinary tract infections, skin/soft tissue infections
3. Admitted and discharged from study site

Patient Exclusion Criteria

1. Subjects >18 years of age
2. Hospital length of stay >7 days
3. Requiring intensive care unit level of care

Parent Inclusion Criteria 1. Parent of eligible child

Parent Exclusion Criteria

1. Parent of ineligible child

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1131 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of suboptimal prescribing | up to 3 years
  The primary objective of this study is to determine the impact of a discharge stewardship intervention on antibiotic prescribing and patient outcomes for three common pediatric infection after developing and implementing the intervention across four geographically diverse children's hospitals. Impact will be measured by the rate of suboptimal prescribing (drug, dose, route, and duration) for CAP, UTI, and SSTI across the four hospitals. Suboptimal prescribing will be measured using data collected from the electronic health record. The discharge prescription data (choice and duration) will be compared to the recommended guidelines to determine if the discharge prescription was on or off guideline.

SECONDARY OUTCOMES:
Impact of the discharge stewardship intervention on post-discharge treatment failure | up to 3 years
  Using a quasi-experimental design, the study team will assess the rate and trajectory of post-discharge treatment failure for CAP, UTI, and SSTI via patient report (post-discharge REDCap surveys)
Impact of the discharge stewardship intervention on adverse drug events | up to 3 years
  Using a quasi-experimental design, the study team will assess the rate and trajectory of adverse drug events for CAP, UTI, and SSTI via patient report (post-discharge REDCap surveys)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gerber, MD, PhD, Principal Investigator — Associate Professor, Pediatrics
Locations (5):
- United States (5):
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
This study was initiated prior to the NIH Data Management and Sharing Policy update that was released on January 25, 2023.

REFERENCES:
- [Background] Hurst AL, Child J, Pearce K, Palmer C, Todd JK, Parker SK. Handshake Stewardship: A Highly Effective Rounding-based Antimicrobial Optimization Service. Pediatr Infect Dis J. 2016 Oct;35(10):1104-10. doi: 10.1097/INF.0000000000001245. PMID 27254036
- [Background] Newland JG, Stach LM, De Lurgio SA, Hedican E, Yu D, Herigon JC, Prasad PA, Jackson MA, Myers AL, Zaoutis TE. Impact of a Prospective-Audit-With-Feedback Antimicrobial Stewardship Program at a Children's Hospital. J Pediatric Infect Dis Soc. 2012 Sep;1(3):179-86. doi: 10.1093/jpids/pis054. Epub 2012 Jul 12. PMID 26619405
- [Background] Gerber JS, Prasad PA, Fiks AG, Localio AR, Grundmeier RW, Bell LM, Wasserman RC, Keren R, Zaoutis TE. Effect of an outpatient antimicrobial stewardship intervention on broad-spectrum antibiotic prescribing by primary care pediatricians: a randomized trial. JAMA. 2013 Jun 12;309(22):2345-52. doi: 10.1001/jama.2013.6287. PMID 23757082
- [Background] Lovegrove MC, Geller AI, Fleming-Dutra KE, Shehab N, Sapiano MRP, Budnitz DS. US Emergency Department Visits for Adverse Drug Events From Antibiotics in Children, 2011-2015. J Pediatric Infect Dis Soc. 2019 Nov 6;8(5):384-391. doi: 10.1093/jpids/piy066. PMID 30137509
- [Background] Gerber JS, Ross RK, Bryan M, Localio AR, Szymczak JE, Wasserman R, Barkman D, Odeniyi F, Conaboy K, Bell L, Zaoutis TE, Fiks AG. Association of Broad- vs Narrow-Spectrum Antibiotics With Treatment Failure, Adverse Events, and Quality of Life in Children With Acute Respiratory Tract Infections. JAMA. 2017 Dec 19;318(23):2325-2336. doi: 10.1001/jama.2017.18715. PMID 29260224
- [Background] Hersh AL, Newland JG, Gerber JS. Pediatric Antimicrobial Discharge Stewardship: An Unmet Need. JAMA Pediatr. 2016 Mar;170(3):191-2. doi: 10.1001/jamapediatrics.2015.3369. No abstract available. PMID 26752682
- [Background] Olson J, Thorell EA, Hersh AL. Evaluation of Discharge Antibiotic Prescribing at a Freestanding Children's Hospital: Opportunities for Stewardship. J Pediatric Infect Dis Soc. 2019 Dec 27;8(6):563-566. doi: 10.1093/jpids/piy127. PMID 30544150
- [Background] Yogo N, Haas MK, Knepper BC, Burman WJ, Mehler PS, Jenkins TC. Antibiotic prescribing at the transition from hospitalization to discharge: a target for antibiotic stewardship. Infect Control Hosp Epidemiol. 2015 Apr;36(4):474-8. doi: 10.1017/ice.2014.85. PMID 25782905
- [Background] Scarpato SJ, Timko DR, Cluzet VC, Dougherty JP, Nunez JJ, Fishman NO, Hamilton KW; CDC Prevention Epicenters Program. An Evaluation of Antibiotic Prescribing Practices Upon Hospital Discharge. Infect Control Hosp Epidemiol. 2017 Mar;38(3):353-355. doi: 10.1017/ice.2016.276. Epub 2016 Nov 28. PMID 27890038
- [Background] Chavada R, Davey J, O'Connor L, Tong D. 'Careful goodbye at the door': is there role for antimicrobial stewardship interventions for antimicrobial therapy prescribed on hospital discharge? BMC Infect Dis. 2018 May 16;18(1):225. doi: 10.1186/s12879-018-3147-0. PMID 29769028
- [Background] Olson SC, Smith S, Weissman SJ, Kronman MP. Adverse Events in Pediatric Patients Receiving Long-Term Outpatient Antimicrobials. J Pediatric Infect Dis Soc. 2015 Jun;4(2):119-25. doi: 10.1093/jpids/piu037. Epub 2014 Apr 30. PMID 26407410
- [Background] Gerber JS, Kronman MP, Ross RK, Hersh AL, Newland JG, Metjian TA, Zaoutis TE. Identifying targets for antimicrobial stewardship in children's hospitals. Infect Control Hosp Epidemiol. 2013 Dec;34(12):1252-8. doi: 10.1086/673982. Epub 2013 Oct 24. PMID 24225609
- [Background] Caplinger C, Crane K, Wilkin M, Bohan J, Remington R, Madaras-Kelly K. Evaluation of a protocol to optimize duration of pneumonia therapy at hospital discharge. Am J Health Syst Pharm. 2016 Dec 15;73(24):2043-2054. doi: 10.2146/ajhp160011. Epub 2016 Nov 2. PMID 27806937
- [Background] Yogo N, Shihadeh K, Young H, Calcaterra SL, Knepper BC, Burman WJ, Mehler PS, Jenkins TC. Intervention to Reduce Broad-Spectrum Antibiotics and Treatment Durations Prescribed at the Time of Hospital Discharge: A Novel Stewardship Approach. Infect Control Hosp Epidemiol. 2017 May;38(5):534-541. doi: 10.1017/ice.2017.10. Epub 2017 Mar 6. PMID 28260538
- [Background] Laible BR, Nazir J, Assimacopoulos AP, Schut J. Implementation of a pharmacist-led antimicrobial management team in a community teaching hospital: use of pharmacy residents and pharmacy students in a prospective audit and feedback approach. J Pharm Pract. 2010 Dec;23(6):531-5. doi: 10.1177/0897190009358775. Epub 2010 Mar 31. PMID 21507858
- [Background] Thampi N, Shah PS, Nelson S, Agarwal A, Steinberg M, Diambomba Y, Morris AM. Prospective audit and feedback on antibiotic use in neonatal intensive care: a retrospective cohort study. BMC Pediatr. 2019 Apr 11;19(1):105. doi: 10.1186/s12887-019-1481-z. PMID 30975119
- [Background] Brehaut JC, Colquhoun HL, Eva KW, Carroll K, Sales A, Michie S, Ivers N, Grimshaw JM. Practice Feedback Interventions: 15 Suggestions for Optimizing Effectiveness. Ann Intern Med. 2016 Mar 15;164(6):435-41. doi: 10.7326/M15-2248. Epub 2016 Feb 23. PMID 26903136
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Background] Charani E, Ahmad R, Rawson TM, Castro-Sanchez E, Tarrant C, Holmes AH. The Differences in Antibiotic Decision-making Between Acute Surgical and Acute Medical Teams: An Ethnographic Study of Culture and Team Dynamics. Clin Infect Dis. 2019 Jun 18;69(1):12-20. doi: 10.1093/cid/ciy844. PMID 30445453
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] Szymczak, J.E. and J. Newland (2018) "The Social Determinants of Antimicrobial Prescribing: Implications for Antimicrobial Stewardship." In: Barlam, TF, MM Neuhauser, PD Tamma and K. Trivedi, eds. Practical Implementation of an Antimicrobial Stewardship Program. Cambridge, UK: Cambridge University Press. Chapter 3

DOCUMENTS (2):
  • Informed Consent Form: Patient Consent (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT05826873/ICF_000.pdf
  • Informed Consent Form: Clinician Verbal Consent (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT05826873/ICF_001.pdf